CLINICAL TRIAL: NCT04503070
Title: The Kinetic and Kinematic Profile of the Upper Extremity During Progressive Phases of the Baseball Swing
Brief Title: Motion Capture: Baseball Swing
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Patrick McCulloch,MD, Principal Investigator, The Methodist Hospital Research Institute
Other Study IDs: Pro00020389
Record Dates: First submitted 2020-08-03; First posted 2020-08-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-08

CONDITIONS: Elbow Force

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Baseball Batters: Participants must be healthy volunteers who accept all provisions of the study and agree to complete the program in its entirety. Participants should have their own bat and relative experience of at least 2 years of hitting a baseball. Ages accepted will be 16-40.
  Interventions: Behavioral: Motion capture participant

INTERVENTIONS:
Behavioral: Motion capture participant — Once participants have undergone appropriate calibration processes, they will perform listed swing progressions:
  1. 15 dry swings with a wiffle bat at low, medium and high effort
  2. 15 dry swings with a weighted bat at low, medium and high effort
  3. 15 swings off of a tee at low, medium and high effort
  4. 15 swings at an underhand toss at low, medium and high effort
  5. 15 swings from a pitching machine at low, medium and high effort

SUMMARY:
The aim of this study will be to assess kinetic and kinematic data during different phases of baseball hitting progressions commonly employed in the rehabilitation setting.

DETAILED DESCRIPTION:
Study participants will undergo consent and history process. Subjects must meet inclusion and exclusion criteria prior to consent. Once consent is obtained, each subject will undergo instruction and training expectations of each swing phase. Once an adequate determination of proficiency has been met, each subject will undergo EMG and MOTUS sleeve placement on each upper extremity:

* Forearm flexors
* Forearm extensors
* Medial epicondyle
* Lateral epicondyle
* Posterior rotator cuff musculature

Once participants have undergone appropriate calibration processes, they will perform listed swing progressions in a randomized order:

A. Dry swings - reduced weight (wiffleball) bat - 5 swings light intensity (25-50% effort), 5 swings moderate intensity (50-75% effort), 5 swings high intensity (75-100% effort) B. Dry swings - normal weight bat - 5 swings light intensity (25-50% effort), 5 swings moderate intensity (50-75% effort), 5 swings high intensity (75-100% effort) C. Tee hitting - normal weight bat - middle strike zone level - 5 swings light intensity (25-50% effort), 5 swings moderate intensity (50-75% effort), 5 swings high intensity (75-100% effort) D. Soft toss - underhand toss from assistant - middle strike zone placement - 5 swings light intensity (25-50% effort), 5 swings moderate intensity (50-75% effort), 5 swings high intensity (75-100% effort) E. Simulated hitting - pitching machine - randomized strike zone placement - 5 swings light intensity (25-50% effort), 5 swings moderate intensity (50-75% effort), 5 swings high intensity (75-100% effort)

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy volunteers who accept all provisions of the study and agree to complete the program in its entirety. Participants should have their own bat and relative experience of at least 2 years of hitting a baseball. Ages accepted will be 16-40.

Exclusion Criteria:

1. Previous history of upper extremity injury
2. Current painful dysfunction resulting in exercise or participation limitation
3. Any health-related exercise limitation as ordered by physician
4. Ages outside of 16-40
5. Inability to access clinic and equipment
6. Inexperience with baseball hitting or inability to follow instructions from study staff.

Ages: 16 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Collegiate baseball players
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2019-10-28 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-01 (Actual)

PRIMARY OUTCOMES:
Force on the elbow | January 21 - 27, 2020
  Medial force (Newtons) across the elbow, normalized to the subject's body mass (kg), was calculated (N/kg).

CONTACTS AND LOCATIONS:
Overall Officials: Patrick McCulloch, MD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Hospital, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Posner M, Cameron KL, Wolf JM, Belmont PJ Jr, Owens BD. Epidemiology of Major League Baseball injuries. Am J Sports Med. 2011 Aug;39(8):1676-80. doi: 10.1177/0363546511411700. Epub 2011 Jun 27. PMID 21709023
- [Background] Li X, Zhou H, Williams P, Steele JJ, Nguyen J, Jager M, Coleman S. The epidemiology of single season musculoskeletal injuries in professional baseball. Orthop Rev (Pavia). 2013 Feb 22;5(1):e3. doi: 10.4081/or.2013.e3. Print 2013 Feb 22. PMID 23705061
- [Background] Robinson TW, Corlette J, Collins CL, Comstock RD. Shoulder injuries among US high school athletes, 2005/2006-2011/2012. Pediatrics. 2014 Feb;133(2):272-9. doi: 10.1542/peds.2013-2279. Epub 2014 Jan 13. PMID 24420804
- [Background] Monti R. RETURN TO HITTING: AN INTERVAL HITTING PROGRESSION AND OVERVIEW OF HITTING MECHANICS FOLLOWING INJURY. Int J Sports Phys Ther. 2015 Dec;10(7):1059-73. PMID 26672900
- [Background] Jack RA 2nd, Burn MB, Sochacki KR, McCulloch PC, Lintner DM, Harris JD. Performance and Return to Sport After Tommy John Surgery Among Major League Baseball Position Players. Am J Sports Med. 2018 Jun;46(7):1720-1726. doi: 10.1177/0363546518762397. Epub 2018 Mar 30. PMID 29601208
- [Background] Begly JP, Guss MS, Wolfson TS, Mahure SA, Rokito AS, Jazrawi LM. Performance outcomes after medial ulnar collateral ligament reconstruction in Major League Baseball positional players. J Shoulder Elbow Surg. 2018 Feb;27(2):282-290. doi: 10.1016/j.jse.2017.09.004. PMID 29332665
- [Background] Chang ES, Bishop ME, Baker D, West RV. Interval Throwing and Hitting Programs in Baseball: Biomechanics and Rehabilitation. Am J Orthop (Belle Mead NJ). 2016 Mar-Apr;45(3):157-62. PMID 26991569
- [Background] Wilk KE, Obma P, Simpson CD, Cain EL, Dugas JR, Andrews JR. Shoulder injuries in the overhead athlete. J Orthop Sports Phys Ther. 2009 Feb;39(2):38-54. doi: 10.2519/jospt.2009.2929. PMID 19194026
- [Background] Wilk KE, Hooks TR. Rehabilitation of the throwing athlete: where we are in 2014. Clin Sports Med. 2015 Apr;34(2):247-61. doi: 10.1016/j.csm.2014.12.010. Epub 2015 Jan 28. PMID 25818712
- [Background] Reinold MM, Wilk KE, Reed J, Crenshaw K, Andrews JR. Interval sport programs: guidelines for baseball, tennis, and golf. J Orthop Sports Phys Ther. 2002 Jun;32(6):293-8. doi: 10.2519/jospt.2002.32.6.293. PMID 12061709
- [Background] Wilk KE, Meister K, Andrews JR. Current concepts in the rehabilitation of the overhead throwing athlete. Am J Sports Med. 2002 Jan-Feb;30(1):136-51. doi: 10.1177/03635465020300011201. PMID 11799012
- [Background] Axe M, Hurd W, Snyder-Mackler L. Data-based interval throwing programs for baseball players. Sports Health. 2009 Mar;1(2):145-53. doi: 10.1177/1941738108331198. PMID 23015866
- [Background] Welch CM, Banks SA, Cook FF, Draovitch P. Hitting a baseball: a biomechanical description. J Orthop Sports Phys Ther. 1995 Nov;22(5):193-201. doi: 10.2519/jospt.1995.22.5.193. PMID 8580946
- [Background] Higuchi T, Nagami T, Morohoshi J, Nakata H, Kanosue K. Disturbance in hitting accuracy by professional and collegiate baseball players due to intentional change of target position. Percept Mot Skills. 2013 Apr;116(2):627-39. doi: 10.2466/30.23.25.PMS.116.2.627-639. PMID 24032335
- [Background] Escamilla RF, Fleisig GS, DeRenne C, Taylor MK, Moorman CT 3rd, Imamura R, Barakatt E, Andrews JR. Effects of bat grip on baseball hitting kinematics. J Appl Biomech. 2009 Aug;25(3):203-9. doi: 10.1123/jab.25.3.203. PMID 19827469
- [Background] Dowling B, Fleisig GS. Kinematic comparison of baseball batting off of a tee among various competition levels. Sports Biomech. 2016 Sep;15(3):255-69. doi: 10.1080/14763141.2016.1159320. PMID 27278749
- [Background] Mahure SA, Mollon B, Shamah SD, Kwon YW, Rokito AS. Disproportionate trends in ulnar collateral ligament reconstruction: projections through 2025 and a literature review. J Shoulder Elbow Surg. 2016 Jun;25(6):1005-12. doi: 10.1016/j.jse.2016.02.036. PMID 27197888
- [Background] Erickson BJ, Eno JJ, Mlynarek RA, Altchek DW. An acute ulnar collateral ligament tear in a professional baseball player while batting requiring ulnar collateral ligament reconstruction. J Shoulder Elbow Surg. 2018 Sep;27(9):e279-e282. doi: 10.1016/j.jse.2018.05.040. Epub 2018 Jul 24. No abstract available. PMID 30054241
- [Background] Lightsey HM, Trofa DP, Sonnenfeld JJ, Swindell HW, Makhni EC, Ahmad CS. Rehabilitation Variability After Elbow Ulnar Collateral Ligament Reconstruction. Orthop J Sports Med. 2019 Mar 25;7(3):2325967119833363. doi: 10.1177/2325967119833363. eCollection 2019 Mar. PMID 30937318
- [Background] Redler LH, Degen RM, McDonald LS, Altchek DW, Dines JS. Elbow ulnar collateral ligament injuries in athletes: Can we improve our outcomes? World J Orthop. 2016 Apr 18;7(4):229-43. doi: 10.5312/wjo.v7.i4.229. eCollection 2016 Apr 18. PMID 27114930
- [Background] Wilk KE, Macrina LC, Cain EL, Dugas JR, Andrews JR. Rehabilitation of the Overhead Athlete's Elbow. Sports Health. 2012 Sep;4(5):404-14. doi: 10.1177/1941738112455006. PMID 23016113
- [Background] Ellenbecker TS, Wilk KE, Altchek DW, Andrews JR. Current concepts in rehabilitation following ulnar collateral ligament reconstruction. Sports Health. 2009 Jul;1(4):301-13. doi: 10.1177/1941738109338553. PMID 23015887